CLINICAL TRIAL: NCT07096817
Title: Fundamental Insights Into the Interplay Between Postural Control and Motor Development in Children With DCD: a Synergistic Approach of Functional Evaluations, Neuromechanics and Brain Activity
Brief Title: Effects of a Highly Intensive Balance Therapy Camp in Children With Developmental Coordination Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Katrijn Klingels, Prof. dr., Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21KP09BOF
Record Dates: First submitted 2025-07-11; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Developmental Coordination Disorder
Keywords: "Postural Balance"[Mesh]; "Pediatrics"[Mesh]; Developmental Coordination Disorder; "Motor Skills Disorders"[Mesh]; Postural Control; Rehabilitation; Functional Therapy; Highly intensive therapy; Motor learning; Individual therapy
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Intervention Model Description: pre-post interventional test design with a triple, nontraining baseline and follow-up. After inclusion, participants are followed for six months prior to the intervention using a triple baseline consisting of six months pre-assessment (T1), a three-months pre-assessment (T2) and a pre-interventional assessment, up to two weeks before the intervention (T3). After the camp, patients perform a post-interventional assessment, up to two weeks after the end of the intervention (T4) and a three-month follow-up assessment (T5)
Masking Description: The Kids-BESTest and TGMD-3 performances are videotaped and scored on video by an experienced assessor. Assessors are blinded for the pre-post condition and timing of the assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Individualized balance therapy (with follow-up after and baseline follow-up) (Experimental): The therapy of the children will be given in intensive camps. A total of four camps are organized between April 2023 and August 2024. Each camp consists of six days of therapy, with a total therapy time of 40 hours. The central camp theme is "Circus", due to the attractiveness for children and the link with postural control. The intervention is functional, and divided in six activity categories: jumping, sitting balance, walking and running, circus, individual goals and group activities with focus on social interaction (Table 2). Each category should: 1. partially or fully cover the multisystemic framework of Horak, with the overall program covering the entire framework , 2. be fun and focusing on collaboration rather than competition.
  During three months prior to the intervention (camps), the children are followed up for six months and assessed at three time points. They will keep on following their usual physiotherapy sessions.
  Interventions: Behavioral: Highly intensive individualized balance therapy

INTERVENTIONS:
Behavioral: Highly intensive individualized balance therapy — In the form of a camp with total therapy hours of 40 hours with a central theme of "Circus", children will receive individualized (1 therapist per child) intensive therapy. The intervention is functional, and divided in six activity categories: jumping, sitting balance, walking and running, circus, individual goals and group activities with focus on social interaction. Each category should: 1. partially or fully cover the multisystemic balance framework of Horak, with the overall program covering the entire framework, 2. be fun and focusing on collaboration rather than competition.

SUMMARY:
The main objective of this clinical trial is to investigate the short (immediately after intervention) and medium term (three month) effects of a highly intensive, comprehensive postural control 6-day therapy camp in school-aged children (6 to 12 years) with developmental coordination disorder at different levels of the The International Classification of Functioning, Disability and Health (ICF) framework.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with DCD by a pediatrician, using the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria: (i) motor skill acquisition and performance is at an age-inappropriate level (Criterion A), objectified with the total MABC-2 score at or below the 16th percentile or subscale score at or below the 5th percentile; (ii) the motor skills deficit significantly and persistently interferes with the activities of everyday living (Criterion B), objectified with the DCD Questionnaire 2007 (DCD-Q) ; (iii) Onset of symptoms in early childhood (Criterion C) evaluated by anamnesis with parents; (iv) The motor skills deficits are not better accounted for by any other medical (neurological, intellectual, visual, etc.), neurodevelopmental, psychological, social condition, or cultural background (criterion D), evaluated by a neuromotor examination performed by an acknowledged pediatrician.
* children who have no formal diagnosis are evaluated by the research team using the diagnostic criteria as outlined in the inclusion criteria. In this case, Criterion D is evaluated based on anamnesis and clinical examination. If criterion A, B, C are met and other intellectual, visual or neurological conditions have not been reported, they are included as having "probable" DCD.
* Due to the interventional focus on postural control, children are only included if they score below the 50th percentile for the balance subscale of the MABC-2 and below 80% on the Kids-BESTest total score.
* Due to the high comorbidity rate in children with DCD, such as attention deficit hyperactivity disorder (ADHD), autism spectrum disorder (ASD) and dyslexia, the comorbidities are listed through thorough anamnesis and the Strengths and difficulties questionnaire (SDQ) is used.

Exclusion Criteria:

- not able to follow instructions or cooperate sufficiently due to behavioral problems

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in Balance Evaluation Systems Test (Kids-BESTest) scores | 6 months pre-assessment, 3 months pre-assessment, pre-interventional assessment (up to two weeks before the start of the intervention), post-interventional assessment (up to two weeks after the end of the intervention), 3 months follow-up assessment
  The Kids-BESTest is a standardized performance tool to assess postural control in children aged between 5 and 18 years old. The test has excellent reliability and consists of 36 items divided over 6 domains. Items are scored from 0 (worst performance) to 3 (normal performance) on 4-point Likert scale. Based on the summation of the task scores, the domain and total scores can be calculated and expressed as a percentage (minimum 0 - maximum 100). A higher score means a better balance performance.

SECONDARY OUTCOMES:
Change in scores on the Canadian Occupational Performance Measure (COPM) | pre-interventional assessment (up to two weeks before the start of the intervention), post-interventional assessment (up to two weeks after the end of the intervention), 3 month follow-up assessment
  The COPM is a client-centered outcome measure to determine and evaluate individual treatment goals. Measurement properties are satisfactory to excellent. In a semi-structured interview between therapist and child (over 8 years) or parents (under 8 years) balance-related problems in daily living are determined. After scoring for importance on a 10-point rating scale (minimum 1 - maximum 10), up to 3 self-selected treatment goals are identified. Each goal is self-rated based on the level of performance and satisfaction. In this study the Dutch version is used. Higher scores indicate more satisfaction and better performance.
Change in scores of the Test of Gross Motor Development, 3rd edition (TGMD-3) | 6 months pre-assessment, 3 months pre-assessment, pre-interventional assessment (up to two weeks before the start of the intervention), post-interventional assessment (up to two weeks after the end of the intervention), 3 months follow-up assessment
  The TGMD-3 is a functional process-oriented test to assess fundamental motor skills in children between 3 and 10 years old, with high test-retest reliability and validity. The test consists of 13 fundamental motor skills, subdivided across two subscales: locomotor and object control skills. Each skill is assessed with three to five performance criteria reflecting the developmental stage of the movement pattern. If a criterion is reached a score 1 is given, if not a score 0 is given. Each skill is assessed 2 times. All criterion scores of the two repetitions of each skill is summed up to obtain the domain scores. These raw domain scores are corrected for age and sex to a scaled score per domain (minimum 1 - maximum 20). Afterwards the scaled score for the total score (gross motor index) is calculated. The scaled scores are used for analyses. A higher score means a better motor performance.
Changes muscle activation patterns during balance tasks (measured with surface electromyography): onset latencies | 6 months pre-assessment, pre-interventional assessment (up to two weeks before the start of the intervention), post-interventional assessment (up to two weeks after the end of the intervention), 3 months follow-up assessment
  Surface EMG is a reliable tool that can be used to measure muscle activity in lumbar and lower limb muscles. Muscle activity is registered using sEMG TrignoTM, Delsys Inc., USA. Registered muscles are: m. gastrocnemius medial head, m. tibialis anterior, m. rectus femoris, m. biceps femoris, m. gluteus medius and mm. erector spinae. Outcome measure regarding sEMG is onset latencies (time in ms). Sensor placement and locations are performed in accordance with the SENIAM guidelines. Muscle activity is registered simultaneously with fNIRS during performance of Kids-BESTest tasks.
Changes muscle activation patterns during balance tasks (measured with surface electromyography): time to peak | 6 months pre-assessment, pre-interventional assessment (up to two weeks before the start of the intervention), post-interventional assessment (up to two weeks after the end of the intervention), 3 months follow-up assessment
  Surface EMG is a reliable tool that can be used to measure muscle activity in lumbar and lower limb muscles. Muscle activity is registered using sEMG TrignoTM, Delsys Inc., USA. Registered muscles are: m. gastrocnemius medial head, m. tibialis anterior, m. rectus femoris, m. biceps femoris, m. gluteus medius and mm. erector spinae. Outcome measure regarding sEMG is time to peak activity (time in ms). Sensor placement and locations are performed in accordance with the SENIAM guidelines. Muscle activity is registered simultaneously with fNIRS during performance of Kids-BESTest tasks.
Changes muscle activation patterns during balance tasks (measured with surface electromyography): co-contraction | 6 months pre-assessment, pre-interventional assessment (up to two weeks before the start of the intervention), post-interventional assessment (up to two weeks after the end of the intervention), 3 months follow-up assessment
  Surface EMG is a reliable tool that can be used to measure muscle activity in lumbar and lower limb muscles. Muscle activity is registered using sEMG TrignoTM, Delsys Inc., USA. Registered muscles are: m. gastrocnemius medial head, m. tibialis anterior, m. rectus femoris, m. biceps femoris, m. gluteus medius and mm. erector spinae. Outcome measure regarding sEMG is co-contraction (percentage). Sensor placement and locations are performed in accordance with the SENIAM guidelines. Muscle activity is registered simultaneously with fNIRS during performance of Kids-BESTest tasks.
Changes in oxy-hemoglobin levels in different cortical brain regions during balance tasks (measured with functional Near-Infrared Spectroscopy) | 6 months pre-assessment, pre-interventional assessment (up to two weeks before the start of the intervention), post-interventional assessment (up to two weeks after the end of the intervention)
  To register cortical brain activity, fNIRS is applied simultaneously with preselected Kids-BESTest tasks. This optical neuro-imaging technique uses infrared light to monitor changes in the concentration (μmol/l) of oxygenated (HbO2) between the task and baseline condition. It is a reliable tool for within-subject measurements and can be reliably applied in children. Due to its portability, it can be used during postural control tasks and gait measurements. The NIRSport 2 (NIRx Medical Technologies, GE) with continuous wave (760nm; 850nm) imaging is used. The region of interests (ROI) targeted with fNIRS were determined based on evidence of brain areas responsible for adequate postural control tasks in healthy individuals and affected brain areas in children with DCD in a variety of tasks. The ROI include the inferior (IPL) and superior parietal lobe (SPL), premotor cortex (PMC) and the supplementary motor area (SMA).
Changes in deoxy-hemoglobin levels in different cortical brain regions during balance tasks (measured with functional Near-Infrared Spectroscopy) | 6 months pre-assessment, pre-interventional assessment (up to two weeks before the start of the intervention), post-interventional assessment (up to two weeks after the end of the intervention)
  To register cortical brain activity, fNIRS is applied simultaneously with preselected Kids-BESTest tasks. This optical neuro-imaging technique uses infrared light to monitor changes in the concentration (μmol/l) of deoxygenated hemoglobin (HHb) between the task and baseline condition. It is a reliable tool for within-subject measurements and can be reliably applied in children. Due to its portability, it can be used during postural control tasks and gait measurements. The NIRSport 2 (NIRx Medical Technologies, GE) with continuous wave (760nm; 850nm) imaging is used. The region of interests (ROI) targeted with fNIRS were determined based on evidence of brain areas responsible for adequate postural control tasks in healthy individuals and affected brain areas in children with DCD in a variety of tasks. The ROI include the inferior (IPL) and superior parietal lobe (SPL), premotor cortex (PMC) and the supplementary motor area (SMA).
Self-perceived competence measured with "Competentiebelevingsschaal voor kinderen (CBSK) (=Dutch) | 6 months pre-assessment, 3 months pre-assessment, pre-interventional assessment (up to two weeks before the start of the intervention), post-interventional assessment (up to two weeks after the end of the intervention), 3 months follow-up assessment
  In children 8-12 years self-perceived competence is assessed with CBSK. The CBSK is reliable and consists of 36 items across six domains: scholastic competence, social acceptation, athletic competence, physical appearance, behavioral conduct and global self-worth. Each item is scored on a 4-point ordinal scale. Raw subscale scores are converted to percentile scores (minimum 0 - maximum 100).
Parents' perception of their child using a qualitative questionnaire and interview parents | pre-interventional assessment (up to two weeks before the start of the intervention), post-interventional assessment (up to two weeks after the end of the intervention), 3 months follow-up assessment
  Parents' perception of their child is questioned with 14 open questions on the child, parents, family and social contacts. Before intervention, parents list their baseline findings, changes are questioned after intervention. Based on these answers, a focus group with the parents is organized at follow-up.
Questionnaire for therapists | pre-interventional assessment (up to two weeks before the start of the intervention), 3 months follow-up assessment
  Details (goals, frequency, duration) on the participants' therapy and potential changes in content since the first baseline measurement were questioned with the therapists before intervention. If during the therapy time before and after the camp, postural control goals were set, training methods were inventoried. On follow-up, changes in therapy goals and potential changes in performance are questioned.
Pictorial scale of perceived competence and social acceptance (PSPCSA) | 6 months pre-assessment, 3 months pre-assessment, pre-interventional assessment (up to two weeks before the start of the intervention), post-interventional assessment (up to two weeks after the end of the intervention), 3 months follow-up assessment
  In children aged 6-7 years, the PSPCSA is used. The PSPCSA is reliable and consists 24 items across 4 domains (cognitive competence, physical competence, peer acceptance and maternal acceptance). Items are scored on a 4-point ordinal scale. Raw subscale scores can be calculated, with higher scores indicating higher competence (minimum 24 - maximum 48).

CONTACTS AND LOCATIONS:
Locations (1):
- Hasselt University, Diepenbeek, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: After publication of results
Access Criteria: Researchers who provide a methodologically sound proposal

REFERENCES:
- [Background] Velghe S, Rameckers E, Meyns P, Johnson C, Hallemans A, Verbecque E, Klingels K. Effects of a highly intensive balance therapy camp in children with developmental coordination disorder - An intervention protocol. Res Dev Disabil. 2024 Apr;147:104694. doi: 10.1016/j.ridd.2024.104694. Epub 2024 Feb 20. PMID 38382234
- See also: website with study information and possibility for enrolment, target group: parents and therapists — https://www.uhasselt.be/nl/onderzoeksgroepen/reval/dcd